CLINICAL TRIAL: NCT00850564
Title: Effect of Short Term Growth Hormone Releasing Hormone in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Steven K. Grinspoon, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK63639B; R01DK063639 (NIH)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2011-03-30 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Volunteers
Keywords: growth hormone releasing hormone
MeSH Terms: interventions — Growth Hormone-Releasing Hormone; tesamorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Hormone Releasing Hormone (Experimental): Growth Hormone Releasing Hormone (Tesamorelin) 2mg by subcutaneous injection once daily
  Interventions: Drug: Growth Hormone Releasing Hormone (Tesamorelin)

INTERVENTIONS:
Drug: Growth Hormone Releasing Hormone (Tesamorelin) — Tesamorelin 2mg subcutaneous daily x 2 weeks
  Other Names: Tesamorelin

SUMMARY:
The purpose of this trial is to examine the short-term effects of Growth Hormone Releasing Hormone (GHRH, tesamorelin) administration in healthy men. We hypothesize that GHRH will increase GH pulse height and will not affect insulin sensitivity.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effects of growth hormone releasing hormone (Tesamorelin) on endogenous overnight growth hormone secretion and pulsatility, as well as insulin-stimulated glucose uptake. Healthy male subjects will receive 2mg Tesamorelin, subcutaneously, daily for two weeks. At baseline and after two weeks of treatment, we will assess overnight growth hormone by frequent sampling as well as insulin stimulated glucose uptake by clamp. Subjects will then stop the Tesamorelin and will return for an identical assessment after a 2 week withdrawal period.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-60 years
* BMI > 20kg/m2 and <35kg/m2

Exclusion Criteria:

* Use of anti-diabetic agents, Megace, testosterone or any steroid use within 6 months of the study
* Use of GH or growth hormone stimulating peptides within six months of starting the study
* Change in lipid lowering or antihypertensive regimen within 3 months of screening
* Fasting blood sugar > 126 mg/dL, SGOT > 2.5 times ULN, Hgb < 12.0 g/dL, creatinine > 1.4 mg/dL
* Carpal tunnel syndrome
* Severe chronic illness or active malignancy or history of pituitary malignancy or history of colon cancer
* For men, history of prostate cancer or evidence of prostate malignancy by PSA > 5 ng/mL
* Prior history of hypopituitarism, head irradiation or any other condition known to affect the GH axis
* Weight < 110 lbs.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Result] Stanley TL, Chen CY, Branch KL, Makimura H, Grinspoon SK. Effects of a growth hormone-releasing hormone analog on endogenous GH pulsatility and insulin sensitivity in healthy men. J Clin Endocrinol Metab. 2011 Jan;96(1):150-8. doi: 10.1210/jc.2010-1587. Epub 2010 Oct 13. PMID 20943777
- [Derived] Makimura H, Stanley TL, Chen CY, Branch KL, Grinspoon SK. Relationship of adiponectin to endogenous GH pulse secretion parameters in response to stimulation with a growth hormone releasing factor. Growth Horm IGF Res. 2011 Jun;21(3):155-9. doi: 10.1016/j.ghir.2011.03.009. Epub 2011 Apr 30. PMID 21531600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment from March 2009 through March 2010
Groups:
- Growth Hormone Releasing Hormone (Tesamorelin): Growth Hormone Releasing Hormone (Tesamorelin) 2mg by subcutaneous injection once daily
Period: Overall Study
Arm/Group | Growth Hormone Releasing Hormone (Tesamorelin)
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Growth Hormone Releasing Hormone (Tesamorelin)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Overnight Growth Hormone
Description: Outcome is mean overnight growth hormone at 2 weeks (i.e., following 2 weeks of treatment with growth hormone releasing hormone). Growth hormone was measured overnight (from 8pm-7:40am) by frequent blood sampling, and the mean is the average of these frequent measurements. The mean measurement at 2 weeks is given here, and, in the statistics section, is statistically compared with the mean measurement before treatment.
Time Frame: at 2 weeks (i.e., after 2 weeks of treatment)
Population: analysis of 13 participants who completed both baseline and 2 week visits
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | Growth Hormone Releasing Hormone (Tesamorelin)
Number analyzed (Participants) | 13
mcg/L | 1.2 (0.3)
Statistical Analysis 1: Comparison: Growth Hormone Releasing Hormone (Tesamorelin); Paired t-test comparing baseline and 2 week mean overnight growth hormone; Test type: Superiority or Other; p < 0.005, Paired t-test

2. Secondary Outcome: Insulin Stimulated Glucose Utilization
Description: Insulin stimulated glucose uptake (M) is the amount of glucose (measured in mg per kg body weight per minute) taken up during the steady state period of a euglycemic hyperinsulinemic clamp. This measure was calculated for minutes 100-120 of euglycemic hyperinsulinemic clamp procedure at 2 weeks (i.e., after 2 weeks treatment with growth hormone releasing hormone). The measurement at 2 weeks is given here, and, in the statistics section, is statistically compared with the measurement before treatment.
Time Frame: at 2 weeks (i.e., after 2 weeks of treatment)
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Growth Hormone Releasing Hormone (Tesamorelin)
Number analyzed (Participants) | 13
mg/kg/min | 7.5 (1.2)
Statistical Analysis 1: Comparison: Growth Hormone Releasing Hormone (Tesamorelin); Paired t-test comparing insulin stimulated glucose uptake (M) between baseline and 2 week visits; Test type: Superiority or Other; p = 0.61, Paired t-test

ADVERSE EVENTS:
Time Frame: Total of 4 weeks: 2 weeks of treatment with study drug, followed by 2 weeks off drug
Description: Subjects queried about potential side effects at 2 week visit (after 2 weeks on study drug) and at 4 week visit (after 2 weeks off drug)
Arm/Group | Growth Hormone Releasing Hormone (Tesamorelin)
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone Releasing Hormone (Tesamorelin) (N=13)
Influenza due to Influenza A virus (Infections and infestations) | 1 (1) — Influenza infection requiring hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone Releasing Hormone (Tesamorelin) (N=13)
chest pain (Cardiac disorders) | 1 (1) — mild chest pain - EKG, cardiac enzymes, stress test all normal.
rash (Skin and subcutaneous tissue disorders) | 1 (1) — mild rash on dorsum of hands, self-resolved
Diarrhea (Gastrointestinal disorders) | 1 (2) — 2 episodes of watery diarrhea, self-resolved
Headache (Nervous system disorders) | 1 (2) — 2 mild headaches, self-resolved
Complaining of itching (Skin and subcutaneous tissue disorders) | 1 (1) — itching and mild swelling around site of intravenous (IV) catheter, self-resolved
Dizziness (Nervous system disorders) | 1 (1) — mild dizziness some mornings while on study medication, resolved on discontinuation
Burn of back (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less